CLINICAL TRIAL: NCT01320046
Title: Vulvar Contact Dermatitis Resulting From Urine Incontinence: Prevalence, Characteristics and Risk Factors
Brief Title: Vulvar Contact Dermatitis Resulting From Urine Incontinence
Status: Withdrawn | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC11029-2011kCTIL
Record Dates: First submitted 2011-03-20; First posted 2011-03-22 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2012-04

CONDITIONS: Urinary Incontinence; Vulvar Pruritus; Vulvar Contact Dermatitis
Keywords: Urinary Incontinence; Vulvar pruritus; Vulvar contact dermatitis
MeSH Terms: conditions — Urinary Incontinence; Pruritus Vulvae | interventions — Surveys and Questionnaires; Vaginal Smears

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal smears taken for evaluation of vaginal estrogen status (identifying parabasal cells, vaginal flora, vaginal pH)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with urinary incontinence: Patients attending the urogynecological clinic for urinary incontinence-100 patients. In this group we will recruit patients with UI, and will assess co-existence of VCD
  Interventions: Other: Questionnaires, gynecological exam , vaginal smear, and measurement of urine leakage
- Patients with vulvar contact dermatitis: Patients attending the vulvovaginal clinic with vulvar contact dermatitis (100 patients). In this group we will recruit patients with VCD, and will assess co-existence of UI.
  Interventions: Other: Questionnaires, gynecological exam , vaginal smear, and measurement of urine leakage
- Age matched control group: Patients attending the general clinic for annual checkup, which will be matched for age with the two other groups (200 patients).
  These patients will be evaluated for symptoms of UI and VCD

INTERVENTIONS:
Other: Questionnaires, gynecological exam , vaginal smear, and measurement of urine leakage — Patients will undergo the following evaluation:
  1. Questionnaires- age, medical background, BMI, UI characteristics , usage of pads, other hygiene practices,hormonal therapy, presence of allergic tendency and history etc.
  2. Medical history.
  3. Gynecological exam including bladder/rectum/uterine prolapse, vaginal atrophy, discharge, findings of VCD (as part of the usual evaluation in the clinic).
  4. Vaginal smear: this will be used for vaginal pH measurement and for wet mount, which will assess estrogen deficiency, yeast infection and other inflammatory conditions. Vaginal smears are done as part of the usual evaluation in the clinic.
  5. Evaluation of the severity of urinary incontinence will be done by collection and weighting of pads during 24 hours.
  Groups: Patients with urinary incontinence; Patients with vulvar contact dermatitis

SUMMARY:
Vulvar contact dermatitis (VCD) is a common problem presenting as vulvar pruritus, burning or irritation. Its estimated prevalence is 20-30% in vulvar clinics, but the prevalence in the general population is unknown.

Contact dermatitis is an inflammation of the skin resulting from an external agent that acts as an irritant or as an allergen. The skin reaction may be acute, subacute or chronic, resulting from prolonged exposure to weak irritating substances.

The most common form of VCD is irritant contact dermatitis, and it usually presents as vulvar itch. The causes that contribute to VCD are increased sensitivity of the vulvar skin to irritants compared to other body parts, decrease in the skin barrier function due to exposure to sweat, urine and vaginal discharge and constant friction of the vulvar area. In menopausal women, lack of estrogen contributes to tissue atrophy and thinning, and may increase the effect of irritants on the vulvar skin.

One of the most common irritating substances that cause VCD is urine. The phenomenon of urine-induced VCD is known as" diaper rash" in babies, and it was also described in bedridden patients using diapers constantly. Women with urine incontinence (UI), a problem that its prevalence in women increases with aging, may use constantly panty liners or pads to prevent urine leakage. The urine is being absorbed in the pad, and the vulvar skin is continually exposed to urine. This can cause VCD, similar to diaper rash. The prevalence of this phenomenon in the general population is unknown.

The patients complain of itch, burning or irritation of the vulvar skin, and on exam erythema, edema and irritated skin are found. As most patients do not connect between UI to their vulvar disorder, and as most care-givers do not ask routinely about UI, the vulvar symptoms are mistakenly attributed to yeast infection or other factors. As the cause to the vulvar complaints is not recognized, patients do not receive proper treatment that requires primary management of UI.

The aim of the study is to evaluate the prevalence of VCD in women with UI and to recognize risk factors for UI induced VCD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of vulvar contact dermatitis, with or without urinary incontinence; OR
* Patients with a diagnosis of urinary incontinence, with or without VCD; OR
* Patients without either UI or VCD, age-matched

Exclusion Criteria:

* Diagnosis of other dermatoses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The prevalence of UI induced VCD will be evaluated in 3 groups:
  1. Patients attending the urogynecological clinic for urinary incontinence-100 patients. In this group we will recruit patients with UI, and will assess co-existence of VCD
  2. Patients attending the vulvovaginal clinic with vulvar contact dermatitis (100 patients). In this group we will recruit patients with VCD, and will assess co-existence of UI.
  3. Patients attending the general clinic for annual checkup, which will be matched for age with the two other groups (200 patients).
  These patients will be evaluated for symptoms of UI and VCD
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of vulvar contact dermatitis among patients with urinary incontinence | one year

SECONDARY OUTCOMES:
Risk factors for urinary incontinence induced vulvar contact dermatitis | one year
  Which risk factors contribute to the development of UI induced VCD: estrogen deficiency, allergic predisposition, other medical problems, UI severity etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramat Eshkol Women health center, Clalit health Services, Jerusalem, Israel

REFERENCES:
- [Background] Margesson LJ. Contact dermatitis of the vulva. Dermatol Ther. 2004;17(1):20-7. doi: 10.1111/j.1396-0296.2004.04003.x. PMID 14756887
- [Background] Farage MA, Miller KW, Berardesca E, Maibach HI. Incontinence in the aged: contact dermatitis and other cutaneous consequences. Contact Dermatitis. 2007 Oct;57(4):211-7. doi: 10.1111/j.1600-0536.2007.01199.x. PMID 17868212
- [Background] Crone AM, Stewart EJ, Wojnarowska F, Powell SM. Aetiological factors in vulvar dermatitis. J Eur Acad Dermatol Venereol. 2000 May;14(3):181-6. doi: 10.1046/j.1468-3083.2000.00080.x. PMID 11032061